CLINICAL TRIAL: NCT01527721
Title: Blurring Strength & Aberrometric Changes Following Corneal Cross-linking (CxL) and CXL Combined With Photorefractive Keratectomy (PRK) in Keratoconus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Senior Lecturer of Ophthalmology, Democritus University of Thrace
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2/2012 37
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Keratoconus
Keywords: keratoconus; CxL; CxL combined with t-PRK
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CxL group (Experimental): Volunteers of this group received CxL treatment.
  Interventions: Procedure: Corneal Collagen Cross-Linking (CxL)
- tCxL group (Experimental): Volunteers of this group received CxL combined with t-PRK treatment
  Interventions: Procedure: Corneal Collagen Cross-Linking combined with t-PRK

INTERVENTIONS:
Procedure: Corneal Collagen Cross-Linking (CxL) — The same surgical procedure was applied to all keratoconus patients that included: Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 30 seconds and subsequent de-epithelialization by means of a hockey knife. Following de-epithelialization, a mixture of 0.1% riboflavin in 20% Dextran solution was instilled to the cornea for 30 minutes (2 drops every 2 minutes) prior to the irradiation, until the stroma was completely penetrated and aqueous was stained yellow. The UVA radiation source was UV-XTM Zurich, . Instillation of riboflavin drops (1 drop every 2 minutes) was continued during irradiation, as well, in order to sustain the necessary concentration of the riboflavin. Moreover, balanced salt solution (BSS) was applied every 6 minutes to moisten the cornea.
  Arms: CxL group
Procedure: Corneal Collagen Cross-Linking combined with t-PRK — For tCxL group, the topo-guided PRK preceded the CXL. The epithelium was mechanically removed with a hockey knife and ablation was performed in a 9.0 mm zone with a maximal intended ablation depth of 50μm. No adjuvant Mitomycin-C was applied in any case. For the photorefractive ablation we used the Allegretto Wave 200 Hz (1.0071-1-0.81/1.208 software/ WaveLight AG, Erlangen, Germany) with the T-CAT ablation profile.
  Arms: tCxL group

SUMMARY:
Primary objective of this study was to assess the impact of the two prevalent therapeutic options, CxL and CxL combined with topography-guided photorefractive keratectomy (t-PRK), on both anterior and posterior corneal High order aberations (HOAs).

DETAILED DESCRIPTION:
The Pentacam Classic (Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04) was used for the sake of the study.32 patients with keratoconus were included in the study. Of them, 19 patients underwent CxL treatment (CxL group), while the rest 13 patients underwent CxL combined with t-PRK (tCxL) [tCxL group]. If both eyes were eligible, only one eye was enrolled in the study.Regarding Scheimpflug camera (Pentacam Classic, Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04 ) measurements, acceptable maps had at least 10.0mm of corneal coverage. Moreover, images with extrapolated data in the central 9.0mm zone were excluded.

For both anterior and posterior corneal surfaces, Pentacam-derived HOAs parameters for both pupil diameters of 4mm and 6mm were calculated, as well as the HOA root mean square (RMS)values. Pentacam-derived HOA measurements were obtained one day prior to treatment and then one year post-op.The impact of the surgical technique (either CXL or tCXL) on spherocylindrical error was evaluated by power vector analysis as described before. Furthermore, manifest refractions comprising of sphere (S), cylinder (C) and axis (φ), were converted into three dioptric powers (M, J0 and J45). Moreover, we calculated the overall blurring strength (B) of the spherocylindrical error by measuring the length of the produced vector.

ELIGIBILITY:
Inclusion Criteria:

* progressive keratoconus

Exclusion Criteria:

* glaucoma or suspicion for glaucoma,
* central corneal thickness (CCT) less than 400μm,
* K-readings more than 60D,
* history of herpetic keratitis,
* pregnancy or nursing,
* underlying autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Higher order corneal aberations | 1 year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Thrace (EIT), Alexandroupoli, Greece

REFERENCES:
- [Result] Labiris G, Sideroudi H, Angelonias D, Georgantzoglou K, Kozobolis VP. Impact of corneal cross-linking combined with photorefractive keratectomy on blurring strength. Clin Ophthalmol. 2016 Apr 1;10:571-6. doi: 10.2147/OPTH.S100770. eCollection 2016. PMID 27099464